CLINICAL TRIAL: NCT07399054
Title: Efficacy and Safety of Esomeprazole 40 mg IV in Post-Surgical Patients Admitted to the ICU (EPIC-ICU)
Brief Title: Efficacy and Safety of Esomeprazole 40 mg IV in Post-Surgical Patients Admitted to the ICU
Status: Not yet recruiting | Type: Observational
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Mohan Ramchandani, Consultant Gastroenterology, Asian Institute of Gastroenterology, India
Other Study IDs: EPIC-ICU
Record Dates: First submitted 2025-12-26; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Stress Ulcers; Reflux Episodes
MeSH Terms: conditions — Duodenal Ulcer | interventions — Esomeprazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single Prospective Observational Cohort - Post-surgical ICU Patients: Eligible post-surgical ICU patients will be enrolled into a single prospective observational cohort after providing written informed consent. All patients will receive Esomeprazole 40 mg intravenous as part of routine post-operative ICU care. Gastric pH impedance monitoring, endoscopic evaluations, and clinical assessments will be performed at predefined time points to observe gastric acid control, reflux parameters, safety, and tolerability. No randomization, blinding, or comparator group is involved.
  Interventions: Drug: Esomeprazole

INTERVENTIONS:
Drug: Esomeprazole — Esomeprazole 40 mg IV will be administered following extubation (~12 hours post-surgery) and subsequently at 24-hour intervals (Day 2 and Day 3) as per routine ICU clinical practice. The drug is not assigned for research purposes but is prescribed as standard care. The study will only observe and record gastric pH parameters, reflux episodes, endoscopic findings, safety, and tolerability.

SUMMARY:
Critically ill patients admitted to intensive care units (ICUs) are predisposed to upper gastrointestinal (GI) bleeding secondary to stress-related mucosal damage. The two most significant independent risk factors for stress ulceration and subsequent GI bleeding in this setting are mechanical ventilation and coagulopathy.1,2 Observational data indicate that proton pump inhibitors (PPIs) remain the most frequently employed prophylactic agents in the ICU.3

Comparative studies evaluating the efficacy of PPIs have shown a positive correlation between their pharmacokinetic properties and acid-suppressive activity. Among available PPIs, esomeprazole demonstrates superior pharmacokinetic characteristics, translating into more effective acid control in clinical use.7,8 In fact, one study reported that the area under the curve (AUC) for esomeprazole was nearly twice that of omeprazole at equivalent doses (14), supporting its enhanced acid-suppressive effect and prolonged maintenance of intragastric pH > 4.9

DETAILED DESCRIPTION:
Esomeprazole, a PPI, has demonstrated robust efficacy in the management of gastroesophageal reflux disease (GERD).4 An intravenous (IV) formulation has been developed to facilitate administration in patients for whom oral therapy is not feasible. A study assessed the safety profile after 1 and 4 weeks, as well as the efficacy after 4 weeks of treatment with esomeprazole 40 mg once daily. Their findings indicated that esomeprazole, administered either as an IV bolus, IV infusion, or orally for 1 week followed by 3 weeks of oral dosing, was well tolerated and effectively promoted mucosal healing.5 Similarly, another studyreported significant improvements in symptom control, with mean reductions in heartburn (91.6%), acid regurgitation (96%), belching (96.8%), epigastric pain (88.4%), and dysphagia (84.7%). Based on both investigator and patient global assessments, 89.2% of cases were rated as having an excellent to good therapeutic response.6

Comparative studies evaluating the efficacy of PPIs have shown a positive correlation between their pharmacokinetic properties and acid-suppressive activity. Among available PPIs, esomeprazole demonstrates superior pharmacokinetic characteristics, translating into more effective acid control in clinical use.7,8 In fact, one study reported that the area under the curve (AUC) for esomeprazole was nearly twice that of omeprazole at equivalent doses (14), supporting its enhanced acid-suppressive effect and prolonged maintenance of intragastric pH > 4.9

In view of this evidence, the present study was designed to evaluate the efficacy of IV esomeprazole for intragastric pH control in post-surgical patients admitted to the ICU, as well as to assess its safety and tolerability in this population

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18-75 years admitted to an ICU post-surgery.
* Non-esophagogastric post-surgical patients.
* An anticipated ICU stay for at least 72 hours.
* Willing to provide consent.

Exclusion Criteria:

* Allergy to the study medications or excipients
* Need for enteral feeding
* Estimated survival of <96 hours
* Pregnant and breastfeeding females.
* History of severe thrombocytopenia, coagulopathy, Child-Pugh Class C liver disease, or organ transplant requiring immunosuppressive therapy.
* On other PPIs and/or NSAIDs for last 48 hrs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Proportion of time intragastric pH ≥4 during the 72 hours post dosing | From enrollment to the end of treatment at 72 hours
  Proportion of time intragastric pH ≥4 during the 72 hours post dosing

SECONDARY OUTCOMES:
• To assess the safety and tolerability of IV Esomeprazole in this patient population, including the incidence of stress ulcers and reflux episodes. | From enrollment to the end of treatment at 72 hours
  • Incidence of stress ulcers and reflux episodes with the help of Proportion of time intragastric pH > 5 and > 6 and Mean intragastric pH on days 1, 2, and 3 post dosing (0-24, 0-48, and 48-72 hrs.)

CONTACTS AND LOCATIONS:
Overall Officials: G V RAO, MBBS,MAMS,FRCS, Principal Investigator — Asian Institute Of Gastroenterology Private Limited

IPD SHARING:
Plan to Share IPD: No